CLINICAL TRIAL: NCT02659748
Title: Examining the Effects of Consuming a Diet Comprising of Milk Fat on Metabolic Health Markers
Brief Title: Milk Fat Intake and Metabolic Health Markers
Acronym: DMFMHM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont Medical Center (Other)
Collaborators: Dairy Research Institute (Other); University of Vermont (Other)
Responsible Party: Principal Investigator, Jana Kraft, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CHRMS M14-011; 1195 (Other Grant/Funding Number: Dairy Research Institute)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Insulin Sensitivity; Type 2 Diabetes
Keywords: Bioactive fatty acids; Insulin sensitivity; Diet; Milk fat; Lipid metabolism; Inflammation markers; Fecal microbiota composition
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milk fat (Experimental): A 21-day low-fat (E%) experimental diet including milk fat with macronutrient and fatty acid class profiles differing only in type of fat and, thus, the proportion of single (bioactive) fatty acids.
  Interventions: Dietary Supplement: Milk Fat
- Control Fat (Experimental): A 21-day low-fat experimental diet. Eucaloric diet to Arm #1 with macronutrient and fatty acid class profiles differing only in type of fat and, thus, the proportion of single fatty acids. A control fat is used to replace dairy fats.
  Interventions: Dietary Supplement: Control Fat

INTERVENTIONS:
Dietary Supplement: Milk Fat — Three daily servings of whole yogurt (3.25% fat).
  Arms: Milk fat
Dietary Supplement: Control Fat — Three daily servings of fat-free yogurt supplemented with a control fat.
  Arms: Control Fat

SUMMARY:
This study investigates the effects of bioactive fatty acids in full fat dairy (whole yogurt), on insulin action, calorie needs, blood lipids, immune function, and body composition in normal and overweight male and female volunteers.

DETAILED DESCRIPTION:
Saturated fats impair the action of insulin leading to abnormally high blood sugar levels that are characteristic of diabetes. Since milk fat is high in saturated fat, some experts advise against whole dairy products (e.g., milk and yogurt). However, bioactive fats, such as those which occur in milk fat, may be beneficial in the prevention of diabetes.

Current data provide no compelling evidence that a moderate intake of saturated fat from milk fat increases the risk of diabetes. Milk fat contains a unique variety of bioactive fats, which may be beneficial and may counterbalance the potential negative effects of saturated fat.

The investigators hypothesize that milk fat has favorable effects on metabolic risk markers associated with the metabolic syndrome. Therefore, this study tests the hypothesis that milk-fat intake will:

(i) result in improved insulin sensitivity,

(ii) favorably alter postprandial lipid metabolism, and

(iii) result in lower circulating concentrations of pro-inflammatory markers.

This study recruits 20-24 (total) female and male subjects in a blinded, randomized, crossover design consisting of two experimental diets (3 weeks each arm) based on a DASH-like diet (Dietary Approaches to Stop Hypertension diet) with % Energy (E%): 55 E% of carbohydrate, 15 E% of protein, and 30 E% of fat (9 E% saturated fatty acids (SFA), 15 E% of monounsaturated fatty acids (MUFA), and 6 E% of polyunsaturated fatty acids (PUFA)). One experimental arm contains milk fat and the other diet contains a control fat.

A washout period represents an average US diet (48 E% of carbohydrate, 15 E% of protein and 37 E% of fat, kcal (16 E% of SFA, 14 E% of MUFA, and 7 E% of PUFA) is used to establish a level of normalization of the fatty acid intake among the subjects and to standardize the subject's physiologic state before each experimental diet.

The two experimental diets are constructed to provide three servings of dairy in the form of either 1) regular whole (full-fat, 3.25%) yogurt or 2) fat-free yogurt supplemented with a control fat. The diets are identical in terms of menus, macro- and micronutrients, and fatty acid class composition (E%) with the exception of individual bioactive fatty acids, allowing for the comparison of the bioactive milk fatty acids to non-milk fatty acids.

At the end of each period (initial washout period and each experimental diet) a frequently sampled intravenous glucose tolerance test is performed, blood is taken for fasting lipids (including lipoprotein profile), serum phospholipid fatty acid profiles, and inflammatory markers, and stool is sampled to examine the fecal microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Good general health and not expecting major lifestyle changes while on study
* BMI between 18.5 and 29.9 kg/m2
* Willing to follow the study coordinator's and dietitian's instructions

Exclusion Criteria:

* Subject with any chronic disease, inflammatory disease and previous diagnosis of HIV or hepatitis C
* Subjects with diabetes (type 1 or 2)
* Subjects with insulin resistance
* Subjects who manifest metabolic syndrome based on aggregate clinical signs
* Intolerance to dairy foods
* Use of prescription medication (except oral contraceptives)
* On medically prescribed diets or following a diet
* Taking supplements that could obscure our ability to detect diet effects
* Frequent use of over-the-counter medication
* Habitual use of tobacco or controlled substances such as cannabis
* Low-density lipoprotein cholesterol (LDL-C) or triacylglycerol (TAG) concentrations <5th or >95th percentile for age
* Participation on regular basis in competitive sports or habitual aerobic exercise training, which we will arbitrarily define as consisting of > 3 bouts/wk of aerobic exercise (unable to speak comfortably) for more than 20 min
* Women who are pregnant or lactating or planning to get pregnant
* Allergies or significant food preferences or restrictions that would interfere with diet adherence
* Lifestyle or schedule incompatible with the study protocol
* Psychiatric or behavioral conditions that in the view of the principal investigator may present a safety hazard to the participant or interfere with study participation or the ability to follow the intervention protocol
* Heart condition

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 3 weeks
  Determined via a frequently sampled intravenous glucose tolerance test (FSIVGTT). Serum samples are analyzed in-house (glucose: glucose oxidase method; insulin: ELISA) to be used in Bergman's minimal model analysis. The results will be used to estimate insulin sensitivity.

SECONDARY OUTCOMES:
Blood lipids | 3 weeks
  Plasma samples analyzed by Nuclear magnetic resonance (NMR) spectroscopy and chemical lipid panel for blood lipids (triacylglycerols, cholesterol profile, including lipoprotein subclasses, lipoprotein particle sizes (Lp(a)),
Inflammation markers. | 3 weeks
  Plasma samples analysed using a high-sensitivity, magnetic, Luminex-based performance assay.
Serum phospholipid analysis | 3 weeks
  Serum phospholipid via SPS analyzed by gas chromatography/mass spectrometry (GC-FID).
Bacterial microbiota | 3 weeks
  Fecal samples collected for the analysis of intestinal bacterial composition using next-generation sequencing (Illumina Miseq V 3.1). Bacterial phyla, classes, orders, and families determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Kraft, PhD, Principal Investigator — University of Vermont; Craig L Kien, MD, Principal Investigator — UVM Medical Center
Locations (1):
- Clinical Research Center, University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes